CLINICAL TRIAL: NCT04580563
Title: Prospective Randomized Versus Placebo Study Assessing Efficacy of Plasmatherapy in Septic Shock-induced Coagulopathy: Feasibility Study
Brief Title: Study Assessing Efficacy of Plasmatherapy in Septic Shock-induced Coagulopathy: Feasibility Study
Acronym: PlasmaFaisa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7572
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Septic Shock; Coagulopathy; Disseminated Intravascular Coagulation
Keywords: septic shock; coagulopathy; disseminated intravascular coagulation; - plasmatherapy
MeSH Terms: conditions — Shock, Septic; Hemostatic Disorders; Disseminated Intravascular Coagulation | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive 12 ml/kg of OctaplasLG® at day 1, within the 2 hours after randomization (i.e. within the 8 hours after coagulopathy diagnosis). A new identical dose will be infused at day 2 according to coagulation parameters.
  OctaplasLG® is a donor plasma product, with unique features compared to standard fresh frozen plasma: standardized concentrations of natural pro-/anti-coagulation factors; a standardized volume; pathogen free. OctaplasLG® should reduce the "inflammatory hit" on the endothelium, including the glycocalyx, by having standardized levels of coagulation proteins, which can give more sustainable support to the endothelial regeneration as compared to standard fresh frozen plasma.
  Interventions: Drug: OctaplasLG®
- Control group (Placebo Comparator): The control group will receive 12 ml/kg of placebo (0.9% NaCl) at day 1, within the 2 hours after randomization (i.e. within the 8 hours after coagulopathy diagnosis). A new identical dose will be infused at day 2 according to coagulation parameters.
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: OctaplasLG® — Patient receive 12 ml/kg of OctaplasLG® at day 1, within the 2 hours after randomization (i.e. within the 8 hours after coagulopathy diagnosis). A new identical dose will be infused at day 2 according to coagulation parameters.
  Arms: Experimental group
Drug: 0.9% NaCl — Patient receive 12 ml/kg of placebo (0.9% NaCl) at day 1, within the 2 hours after randomization (i.e. within the 8 hours after coagulopathy diagnosis). A new identical dose will be infused at day 2 according to coagulation parameters.
  Arms: Control group

SUMMARY:
No randomized controlled trial (RCT) has investigated the effect of prophylactic fresh frozen plasma (FFP) transfusion in septic or critically ill patients with coagulation abnormalities. The last Surviving Sepsis Campaign therefore suggests with a very low quality of evidence "against the use of fresh frozen plasma during septic shock to correct clotting abnormalities in the absence of bleeding or planned invasive procedures". However, expert opinion highlights that FFP should be transfused "when there is a documented deficiency of coagulation factors (increased prothrombin time, international normalized ratio - INR, or partial thromboplastin time) and the presence of active bleeding or before surgical or invasive procedures". Disseminated intravascular coagulation (DIC) is responsible for such a severe deficiency of coagulation factors. Supplementing the intense deficit of coagulation factors with plasma containing non-activated coagulation factors is therefore a rational therapy in DIC patients.

OctaplasLG® is a donor plasma product, with unique features compared to standard fresh frozen plasma: standardized concentrations of natural pro-/anti-coagulation factors; a standardized volume; pathogen free. OctaplasLG® should reduce the "inflammatory hit" on the endothelium, including the glycocalyx, by having standardized levels of coagulation proteins, which can give more sustainable support to the endothelial regeneration as compared to standard fresh frozen plasma.

DETAILED DESCRIPTION:
The present RCT is an open-label faisability study. OctaplasLG® or a placebo (0.9% NaCl) will be allocated to patients with a septic shock-induced coagulopathy defined by decreased platelets (<150,000/mm3 or >30% decrease within 24 hours) and an INR>1.40, and started within the 6 hours following coagulopathy diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with:

  * a septic shock defined by Sepsis-3 criteria (Singer, JAMA 2016)
  * and a coagulopathy assessed by decreased platelets (<150,000/mm3 or >30% decrease within 24 hours) and an INR>1.40 (Vincent, Crit Care Med 2013) without other etiology
* Randomization within a timeframe of 6 hours after coagulopathy diagnosis
* Age strictly over 18 years old
* Subject affiliated to a social health insurance
* Free and informed consent dated and signed.

Exclusion Criteria:

* Contraindication to OctaplasLG®
* Contraindication to preventive anticoagulation by heparin
* Any disorder with a requirement for full anticoagulation on the day of randomization
* PT prolongation or thrombocytopenia that is not due to sepsis
* History of congenital bleeding disorder predisposing to hemorrhage
* Medical condition associated with a hypercoagulable state
* Patient moribund on the day of randomization
* Do not resuscitate limitation at inclusion in the study
* Law protection: guardianship or curatorship
* Pregnancy/breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
delays between the diagnosis of coagulopathy and the administration of treatment | Day 2

SECONDARY OUTCOMES:
Mortality | Day 7
SOFA | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Julie HELMS, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No